CLINICAL TRIAL: NCT00642863
Title: Brain and Behavior Depending on Timing of Iron Deficiency in Human Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2P01HD039386-06A1 (NIH); 2P01HD039386-06A1 (NIH)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-03

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
Keywords: iron deficiency; iron deficiency anemia; infant; development; behavior
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Behavior | interventions — ferrous sulfate; Fluid Therapy; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Low birth iron (Experimental): Infants with low birth iron who receive vitamins A and D + iron
  Interventions: Dietary Supplement: Ferrous Sulfate (liquid) + vitamins A and D
- Marginal birth iron 1 (Experimental): Infants with marginal birth iron randomized to receive vitamins A and D + iron
  Interventions: Dietary Supplement: Ferrous Sulfate (liquid) + vitamins A and D
- Marginal birth iron 2 (Active Comparator): Infants with marginal birth iron randomized to receive vitamins A and D without iron
  Interventions: Dietary Supplement: vitamins A and D
- Normal birth iron (Active Comparator): Infants with normal birth iron who receive vitamins A and D without iron
  Interventions: Dietary Supplement: vitamins A and D
- Combined ID (Experimental): Marginal-birth-iron vitamins only-treated infants who have IDA at 9 mo.
  Interventions: Dietary Supplement: Ferrous sulfate (liquid)
- Early postnatal IDA (Experimental): Infants with IDA at 9 months whose cord blood was collected at birth but who were not assessed and assigned to vitamins with or without iron at 6 weeks
  Interventions: Dietary Supplement: Ferrous sulfate (liquid)
- Late postnatal IDA (Experimental): Infants with IDA at 18 months whose cord blood was collected at birth but who were not assessed and assigned to vitamins with or without iron at 6 weeks. These infants were also not anemic when screened at 9 months.
  Interventions: Dietary Supplement: Ferrous sulfate (liquid)

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate (liquid) + vitamins A and D — a single daily dose of 1-2 mg/kg of elemental iron (5 mg from 6 wk to 9 mo and 15 mg from 9 to 18 mo.) and 1500 IU vitamin A and 500 IU vitamin D from 6 wk to 18 mo.
  Arms: Low birth iron; Marginal birth iron 1
Dietary Supplement: vitamins A and D — a single daily dose (liquid) of 1500 IU vitamin A and 500 IU vitamin D from 6 wk to 18 mo.
  Arms: Marginal birth iron 2; Normal birth iron
Dietary Supplement: Ferrous sulfate (liquid) — Infants who become iron deficient/anemic at 9 or 18 mo will take a single daily dose of 3 mg/kg of elemental iron for 3 months.
  Arms: Combined ID; Early postnatal IDA; Late postnatal IDA

SUMMARY:
It is common in many populations that babies develop iron deficiency or iron deficiency anemia (that is, too few healthy red blood cells due to lack of iron). This is due to rapid growth in infancy combined with limited sources of iron in the infant diet. The amount of iron the baby receives across the placenta during pregnancy is another important factor. This study focuses on infants who are born with less than the usual amount of iron in their bodies. The purposes of the study are to assess effects of lower iron at birth on infant behavior and development and to determine if providing iron supplements to such infants beginning at 6 weeks fosters healthier development. Another part of the study will determine the effects of iron deficiency anemia at different times during infant development.

DETAILED DESCRIPTION:
The project focuses on brain-behavior effects depending on the timing of iron deficiency (ID) and iron repletion in human infants. Iron deficiency (ID) is the world's most common single nutrient disorder, differentially affecting pregnant women and infants everywhere. The study promises to be the first systematic investigation of brain and behavior effects of prenatal dietary iron deficiency in human infants. The design will support comparisons of brain/behavior effects depending on the timing and duration of ID. The study will assess reversibility of effects, depending on timing of ID and its treatment, and examine maternal vs. fetal iron regulatory mechanisms in placenta and white blood cells. State-of-the-art neurophysiologic and behavioral measures will test specific hypotheses regarding effects of ID on sensory, motor, cognitive, affective-social and regulatory functions related to impaired myelination of sensory/motor systems and altered structure, neurotransmitter function and neurometabolism in targeted brain regions (basal ganglia and hippocampus). The study will be conducted in China, a rapidly developing country where ID often occurs among pregnant women and infants in the absence of generalized undernutrition. Cord blood hemoglobin (Hb) and ferritin concentrations will be measured in 1300 rural full-term infants, with iron status determined again at 9 and 18 mo. Brain-behavior assessments in the perinatal period will involve 359 infants ("newborn cohort"): 59 with low Hb ("low birth iron" group) will receive iron; 200 with marginal Hb or low cord ferritin ("marginal birth iron" group) will be randomly assigned at 6 wk, 50 to iron therapy and 150 to vitamins only; and 100 with normal cord Hb and ferritin levels ("normal birth iron" group) will receive vitamins only. The remaining 763 infants with cord blood testing will form the "blood screen cohort." At 9 and 18 mo, the newborn cohort will be reassessed, along with IDA infants from the blood screen cohort - about 58 at 9 mo ("early postnatal IDA") and 48 at 18 mo ("late postnatal IDA"). Approximately 39 marginal-birth-iron vitamins only-treated infants in the newborn cohort may also have IDA at 9 mo ("combined ID"). IDA infants will be treated with vitamins with iron. Differential effects and/or reversibility depending on timing of ID or treatment could inform health policy and practice worldwide. However, the effects of prenatal iron deficiency have received very little study in human infants due in large part to previous thinking, no longer accepted, that the infant was protected. Up to 75% of pregnant women worldwide are anemic, with about half due to ID. An estimated 20-25% of 6- to 24-mo-old infants have IDA, and more have ID without anemia. Thus, the public health implications of study findings could be profound.

The project is expected to continue with a 5-year follow-up (Aug 2013-July 2017).

ELIGIBILITY:
Inclusion Criteria:

* infants born at Maternity and Children's Hospitals of Fuyang city in China
* healthy term newborns from uncomplicated pregnancies for hematology screening
* healthy full-term singleton infants with cord Hb and ferritin in the low-marginal or normal range for developmental testing

Exclusion Criteria:

* perinatal complications

Max Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1614 (Actual)
Dates: Start 2008-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Infant behavior and development | 6 weeks; 9 and 18 months

SECONDARY OUTCOMES:
Low or marginal birth iron | 6 weeks
Infant anemia | 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lozoff, MD, Principal Investigator — University of Michigan; Jie Shao, MD, Study Director — Children's Hospital, Zhejiang University School of Medicine; Zhengyan Zhao, MD, Study Director — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Clark KM, Li M, Zhu B, Liang F, Shao J, Zhang Y, Ji C, Zhao Z, Kaciroti N, Lozoff B. Breastfeeding, Mixed, or Formula Feeding at 9 Months of Age and the Prevalence of Iron Deficiency and Iron Deficiency Anemia in Two Cohorts of Infants in China. J Pediatr. 2017 Feb;181:56-61. doi: 10.1016/j.jpeds.2016.10.041. Epub 2016 Nov 8. PMID 27836288